CLINICAL TRIAL: NCT02693665
Title: Building Evidence for Effective Palliative/End of Life Care for Teens With Cancer
Acronym: FACE-TC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maureen Lyon (Other)
Collaborators: St. Jude Children's Research Hospital (Other); Akron Children's Hospital (Other); National Institute of Nursing Research (NINR) (NIH); Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor-Investigator, Maureen Lyon, Maureen E. Lyon, PhD, ABPP, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00005648; 1R01NR015458-01 (NIH)
Record Dates: First submitted 2016-02-17; First posted 2016-02-29 (Estimated); Results first posted 2025-01-14 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Cancer
Keywords: pediatric advance care planning; adolescent; family; palliative care; end of life; communication; decision making; surrogate decision maker; health care proxy; intervention; randomized clinical trial; cancer; quality of life; spiritual; religion; treatment congruence; treatment preferences; FAmily CEntered (FACE) Advance Care Planning
MeSH Terms: conditions — Neoplasms; Death; Communication; Facies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FACE-TC Intervention (Experimental): Adolescent/family dyads randomized to the experimental condition receive Family Centered Advance Care Planning for Teens with Cancer (FACE-TC) intervention - 3 sessions scheduled one week apart of approximately 60 minutes duration each. Session 1 - Lyon Advance Care Planning Survey-Adolescent & Surrogate versions. Session 2 - Respecting Choices Interview facilitated by trained/certified facilitator with adolescent and family. Focuses on patient's understanding of their illness, possible complications, goals of care and treatment preferences in 3 bad outcome situations; and the Session 3 - Five Wishes an advance directive.
  Interventions: Behavioral: FAmily CEntered Advance Care Planning for Teens with Cancer
- Treatment As Usual (TAU) (No Intervention): Adolescent/family dyads randomized to the treatment as usual (TAU) condition receive written information on advance care planning, but no active intervention.

INTERVENTIONS:
Behavioral: FAmily CEntered Advance Care Planning for Teens with Cancer — 3 session weekly intervention: 1) survey completed by adolescent and family (surrogate decision maker) separately with facilitator; 2) Respecting Choices structured interview about patient's representation of illness, goals of care, hopes, treatment preferences; 3) completion of an advance directive.
  Other Names: FACE-TC
  Arms: FACE-TC Intervention

SUMMARY:
To test the efficacy of FACE-TC on key outcomes, the investigators propose using an intent-to-treat, longitudinal, prospective, multi-site, randomized controlled trial (RCT) design. Adolescents with cancer, aged 14 up to 20 years, and their families (N=130 dyads; N=260 participants) will be recruited and randomized to FACE-TC or Treatment as Usual (TAU) control. Participants will complete standardized questionnaires at baseline and 3, 6, 12, and 18 months post-intervention. Our goal is to assess the extent to which FACE-TC helps adolescents and young adults with cancer and their families: (1) reach and maintain better congruence in treatment preferences over time; (2) improve their quality of life; and (3) document goals of care and advance directives earlier in the course of their potentially life limiting illness.

DETAILED DESCRIPTION:
The investigators propose a prospective, longitudinal, 2-arm RCT to test the efficacy of FACE-TC on key measurable outcomes through 18 months post-intervention. Dyads composed of adolescents with cancer and their families (N=130 dyads; 260 subjects) will be enrolled and randomized to either the FACE-TC intervention or Treatment as Usual (TAU) Control group at a ratio of 2:1 [N=87 FACE-TC dyads and N=43 TAU Control dyads]. The investigators estimate 30% attrition by the 18 month post-intervention assessment (20%-25% due to death/complications and 10% due to dropout). Of the original sample of 130 randomized dyads (N=260 subjects), the investigators estimate the investigators will have full longitudinal data at 18 months post-intervention for 91 dyads (N=182 subjects). Participants will be recruited from Akron Children's Hospital, St. Jude Children's Research Hospital and University of Minnesota Masonic Children's Hospital pediatric oncology programs. Participants will undergo written informed consent/assent. Eligible participants will be enrolled and complete the baseline assessment followed by randomization. Randomization will be at the level of the dyad. Allocation will be concealed from the RA-Assessor to prevent bias. Block randomization by study site will control for site differences. Intervention and Control Conditions: The curriculum based FACE-TC consists of: The Session 1 ACP Survey; Session 2 Respecting Choices Interview; and the Session 3 Five Wishes advance directive. To minimize the burden to ill adolescents, the investigators have chosen a Treatment as Usual comparison condition. This group will be provided with an advance care planning booklet/information only. Assessments occur at baseline, and 3, 6, 12, and 18 months post-intervention. At each site the assessments and intervention will be administered by a research team comprised of the site Co-Investigator and two Research Assistants (RA) (RA-Assessor & RA-Interventionist).Visit protocol: Screening Visit: The RA-Assessor presents the adolescent with cancer and family with an Information Sheet describing the study and conduct an initial assessment about whether they are eligible for enrollment. After consent/assent, further screening for inclusion/exclusion criteria is conducted. Baseline Visit: At enrollment and prior to randomization, baseline measures will be obtained. Entry of baseline data by the RA-Assessor will trigger computerized randomization of patient/family dyads to either FACE-TC intervention or TAU Control using a randomly permuted block design and a 2:1 ratio by study site. The Children's National clinical coordinator will then notify the RA-Interventionist who will schedule the next study visit. The adolescent and family will learn their assignment when the RA-Interventionist calls to schedule study sessions. Attendance will be recorded to assess effects of full vs. partial participation in FACE-TC. Follow-up Visits: RA-Assessor will obtain follow-up measures from the adolescent and family at 3, 6, 12 and 18 month post intervention.

Site Co-Is will oversee site activities and provide weekly, face-to-face supervision of the RAs. They are responsible for recruitment, retention, safety, fidelity to protocol, and supervision and support of RAs. The RAs will assist with recruitment, screening, enrollment and baseline screening measure collection, as well as the day-to-day functioning. RAs will be blind to random assignment. RA-Interventionists will be trained to implement the protocol. Only the RA-Assessor will be permitted to administer post-randomization assessments. Children's National will serve as the data coordinating center and will be responsible for database design and maintenance and the statistical analyses. Sites will be overseen by a Safety Monitoring Committee (SMC). A 2-day Investigator Meeting will be held in Washington, District of Columbia (DC) and will include all site Co-Is, RA-Assessors and consultants. The protocol, its scientific rationale, underlying ethics issues, implementation including recruitment and retention, will be reviewed with the entire team. In month 9 of Year 1 there will be a 3-day training meeting of the RA-Interventionists and RA-Assessors on the intervention, which site-Co-Is will also attend. RA-Assessors will attend only one day of this training in order to maintain blindness. Site Initiation. To begin screening/enrollment (1) the protocol must be approved at each site's Institutional Review Board (IRB) and all personnel must be certified in Human Subjects Research training, (2) personnel are recruited and trained for RA roles, and (3) each RA-Interventionist must complete certification as a Next Steps-ACP Facilitator. Dr. Lyon and the Research Coordinator will verify that the site has all components in place for the logistics of screening, enrolling, scheduling, performing assessments, administering interventions, and collecting the data. To assure continuous quality for the intervention and its evaluation, monitoring will be ongoing. Dr. Lyon and Ms. Briggs will review the first 5 DVD/audio recordings of intervention sessions from each site to ensure fidelity with the protocol. Thereafter, they will randomly review 1 DVD per week, rotating sites. Dr. Lyon and Ms. Briggs will use a competency checklist. Dr. Lyon and Research Coordinator will monitor ongoing site IRB approval documentation and assist sites in annual continuing reviews. The Research Coordinator will keep copies of all regulatory forms, including consent-stamped templates from each site and staff members' Human Subjects Research Training approval certificates. Dr. Lyon and the Research Coordinator will perform twice yearly site monitoring visits while the intervention is being implemented to assure standardization of procedures and resolve any problems that are identified. They will review and confirm that all consents have occurred properly at the sites and that the sites are maintaining all participant and regulatory data. The REDCap database from the FACE-TC pilot will be updated and expanded for this study, and the systems for data entry will be revised to address multi-site implementation. A data dictionary will be created. An external Safety Monitoring Committee (SMC) will be assembled by Dr. Lyon with the responsibility of reviewing safety information, study progress, and other relevant data. The SMC will meet a minimum of once a year. Prior to parametric testing, scale reliabilities for multi-item measures (e.g., pain/fatigue, child and parent psychological, spiritual/religious measures) will be assessed using Cronbach's alpha and their composite scores will be used for data analyses. Analytical Plan for AIM 1. To evaluate the efficacy of FACE-TC on adolescent-family congruence in treatment preferences. Congruence in decision-making for medical treatment will be tested based on agreement (i.e., both patient and his/her family choose the same option) on the Statement of Treatment Preferences in four different cancer-related situations. Kappa coefficients will be applied to assess chance-adjusted agreement between patient and family responses. Change in Kappa coefficient (congruence improvement) from baseline to each follow-up time point during the study period will be tested using bootstrapping technique. The latent growth model (LGM) with categorical outcome will be used to test Hypotheses H1a, i.e., FACE-TC participants will have a higher congruence rate over time. In the LGM, the investigators will set time scores, except those for identification purpose, as free parameters to let the shape of growth trajectory be determined by data. As such, the congruence development trajectory would have an empirically based nonlinear shape, instead of assuming a linear or nonlinear polynomial function. The investigators will apply the growth mixture model (GMM) to test heterogeneity of congruence development trajectories and identify possible patterns of congruence in development trajectories in the full sample. The latent class variable estimated from the GMM captures the pattern of congruence development trajectories. Time-invariant covariates will be used to predict the memberships of the latent trajectory groups; and time-varying covariates will be included to predict the level of congruence at different time points. To test Hypotheses H1b, the investigators will regress the latent growth slope factor and the latent class variable on FACE-TC intervention, controlling for covariates in the GMM to assess 1) how FACE-TC would affect the membership of the latent classes of congruence development; and 2) how the effect of FACE-TC on congruence change over time varies across the latent trajectory classes. Analytical Plan for AIM 2. To evaluate efficacy of FACE-TC on AYA quality of life and family QOL. The LGM and GMM models proposed for evaluating Aim 1 can be readily applied to evaluate Aim 2 and test Hypotheses H2 where the outcome measures are continuous variables. When examining the effects of FACE-TC on QOL for AYAs with cancer and their families, socio-demographics will be controlled as time-invariant covariates, while time-varying covariates will be included in the model to predict measures of QOL at different time points. In addition, family caregiver appraisal/depression measured at the end of the study period will be included as a distal outcome in the GMM models, and how this distal outcome is associated with the patterns of the developmental trajectories of AYA QOL will be assessed. As the same model will be used to evaluate multiple outcomes, Bonferroni correction will be applied to exert a stringent control over false discovery. As attrition is inevitable in longitudinal studies, robust model estimator (e.g., MLR) using the full information maximum likelihood will be used for model estimation. Importantly, missing at random (MAR), instead of missing completely at random, can be assumed in MLR. MAR is a plausible assumption that allows missingness to be dependent on observed measures like intervention assignment. Analytical Plan for AIM 3. To evaluate the efficacy of FACE-TC on early completion of pACP goals of care and advance directives. First, the investigators will use the two-proportion z-test to test the differences in proportions of completion of pACP goals of care and advance directives between FACE-TC and control groups. Then logistic regressions will be used to test the Hypothesis H3, controlling for socio-demographics. Interaction between intervention and ethnicity will be included in the models to test ethnic disparity in regard to intervention efficacy. The investigators will also explore if FACE-TC improves the match between patients' goals of care and the medical care received at the EOL among the adolescents who may die. Descriptive statistics will be used to estimate the frequencies of the study variables. Chi-square statistics with Fisher Exact tests will be used to assess the difference in the match between FACE-TC and controls; and exact logistic regression will be applied to examine the effect of FACE-TC on such a match, controlling for covariates. For continuous outcomes with a modest observation autocorrelation (p=0.20) and moderate effect size (delta=0.35), the estimated sample size to achieve a power of 0.80 at =0.05 level and detect a moderate effect size (delta=0.35) is about N=76 individuals at each of the 5 observation time points. For binary outcomes, a sample size of N=70 can achieve a power of 0.80 to detect a moderate response probability difference of d=0.17 given p=0.20. Our proposed sample of N=130 dyads will ensure a large enough statistical power for our proposed longitudinal analyses on patient data and parent data, respectively. For the cross-sectional logistic regression model proposed to evaluate Aim 3, a sample size of N=100 would achieve a power of 0.83 at alpha=0.05 level to detect an odds ratio of 4.

ELIGIBILITY:
AYA Inclusion Criteria:

* Ever diagnosed with cancer;
* Knows his or her cancer status;
* Ages of 14 up to 20 years;
* Ability to speak English;
* Consent from the legal guardian for adolescents aged 14-17;
* Consent from a surrogate for adolescents aged 18-20;
* Assent from adolescent aged 14-17;
* Consent from adolescent aged 18-20;

Inclusion Criteria for Legal Guardians of Adolescents Age 14-17:

* Legal guardian of assenting adolescent participant;
* Knows cancer status of adolescent;
* Adolescent willingness to discuss problems related to cancer with them;
* Age 18 or older;
* Ability to speak English;
* Consent to participate; Consent for his/her adolescent to participate;

Inclusion Criteria for Surrogates of AYAs Age 18-20:

* Selected by adolescent aged 18 to 20;
* Knows cancer status of adolescent;
* Age 18 or older;
* Ability to speak English;
* Willingness to discuss problems related to cancer and EOL;
* Consent to participate;

Exclusion Criteria - for AYA or surrogate decision-maker:

Developmental delay; foster care; active homicidality or suicidality, depression in the severe range

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2016-07-16 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E Lyon, PhD, Principal Investigator — Children's National Research Institute
Locations (4):
- United States (4):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Akron Children's Hospital, Akron, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
No, only de-identified data.
Supporting Information: Study Protocol, SAP
Time Frame: Estimated April 30, 2022
Access Criteria: Graduate students in accredited programs, residents, fellows and faculty from accredited programs.

REFERENCES:
- [Background] Lyon ME, Jacobs S, Briggs L, Cheng YI, Wang J. A longitudinal, randomized, controlled trial of advance care planning for teens with cancer: anxiety, depression, quality of life, advance directives, spirituality. J Adolesc Health. 2014 Jun;54(6):710-7. doi: 10.1016/j.jadohealth.2013.10.206. Epub 2014 Jan 7. PMID 24411819
- [Background] Lyon ME, Jacobs S, Briggs L, Cheng YI, Wang J. Family-centered advance care planning for teens with cancer. JAMA Pediatr. 2013 May;167(5):460-7. doi: 10.1001/jamapediatrics.2013.943. PMID 23479062
- [Background] Lyon ME, Garvie PA, Briggs L, He J, McCarter R, D'Angelo LJ. Development, feasibility, and acceptability of the Family/Adolescent-Centered (FACE) Advance Care Planning intervention for adolescents with HIV. J Palliat Med. 2009 Apr;12(4):363-72. doi: 10.1089/jpm.2008.0261. PMID 19327074
- [Background] Lyon ME, Garvie PA, Briggs L, He J, Malow R, D'Angelo LJ, McCarter R. Is it safe? Talking to teens with HIV/AIDS about death and dying: a 3-month evaluation of Family Centered Advance Care (FACE) planning - anxiety, depression, quality of life. HIV AIDS (Auckl). 2010;2:27-37. doi: 10.2147/hiv.s7507. Epub 2010 Feb 18. PMID 22096382
- [Background] Lyon ME, Garvie PA, McCarter R, Briggs L, He J, D'Angelo LJ. Who will speak for me? Improving end-of-life decision-making for adolescents with HIV and their families. Pediatrics. 2009 Feb;123(2):e199-206. doi: 10.1542/peds.2008-2379. PMID 19171571
- [Background] Jacobs S, Perez J, Cheng YI, Sill A, Wang J, Lyon ME. Adolescent end of life preferences and congruence with their parents' preferences: results of a survey of adolescents with cancer. Pediatr Blood Cancer. 2015 Apr;62(4):710-4. doi: 10.1002/pbc.25358. Epub 2014 Dec 24. PMID 25545105
- [Background] Wilkins ML, Dallas RH, Fanone KE, Lyon ME. Pediatric palliative care for youth with HIV/AIDS: systematic review of the literature. HIV AIDS (Auckl). 2013 Jul 29;5:165-79. doi: 10.2147/HIV.S44275. Print 2013. PMID 23930080
- [Background] Garvie PA, He J, Wang J, D'Angelo LJ, Lyon ME. An exploratory survey of end-of-life attitudes, beliefs, and experiences of adolescents with HIV/AIDS and their families. J Pain Symptom Manage. 2012 Sep;44(3):373-85.e29. doi: 10.1016/j.jpainsymman.2011.09.022. Epub 2012 Jul 7. PMID 22771129
- [Background] Lyon ME, McCabe MA, Patel KM, D'Angelo LJ. What do adolescents want? An exploratory study regarding end-of-life decision-making. J Adolesc Health. 2004 Dec;35(6):529.e1-6. doi: 10.1016/j.jadohealth.2004.02.009. PMID 15581537
- [Background] Rosenberg AR, Wolfe J, Wiener L, Lyon M, Feudtner C. Ethics, Emotions, and the Skills of Talking About Progressing Disease With Terminally Ill Adolescents: A Review. JAMA Pediatr. 2016 Dec 1;170(12):1216-1223. doi: 10.1001/jamapediatrics.2016.2142. PMID 27749945
- [Background] Lyon ME, D'Angelo LJ, Dallas RH, Hinds PS, Garvie PA, Wilkins ML, Garcia A, Briggs L, Flynn PM, Rana SR, Cheng YI, Wang J. A randomized clinical trial of adolescents with HIV/AIDS: pediatric advance care planning. AIDS Care. 2017 Oct;29(10):1287-1296. doi: 10.1080/09540121.2017.1308463. Epub 2017 Mar 30. PMID 28359212
- [Background] Weaver MS, Anderson B, Cole A, Lyon ME. Documentation of Advance Directives and Code Status in Electronic Medical Records to Honor Goals of Care. J Palliat Care. 2020 Oct;35(4):217-220. doi: 10.1177/0825859719860129. Epub 2019 Jul 7. PMID 31280659
- [Background] Feudtner C, Rosenberg AR, Boss RD, Wiener L, Lyon ME, Hinds PS, Bluebond-Langner M, Wolfe J. Challenges and Priorities for Pediatric Palliative Care Research in the U.S. and Similar Practice Settings: Report From a Pediatric Palliative Care Research Network Workshop. J Pain Symptom Manage. 2019 Nov;58(5):909-917.e3. doi: 10.1016/j.jpainsymman.2019.08.011. Epub 2019 Aug 21. PMID 31445136
- [Background] Watson A, Weaver M, Jacobs S, Lyon ME. Interdisciplinary Communication: Documentation of Advance Care Planning and End-of-Life Care in Adolescents and Young Adults With Cancer. J Hosp Palliat Nurs. 2019 Jun;21(3):215-222. doi: 10.1097/NJH.0000000000000512. PMID 30829829
- [Background] Needle J, Brunnquel D, Lyon M. Mature minors, mature decisions: Advance care planning for adolescent patients with life-limiting illness. Journal of Pediatric Ethics! Advanced Care Planning and End of Life. 2018;1(3).
- [Background] Weaver MS, Bell CJ, Diver JL, Jacobs S, Lyon ME, Mooney-Doyle K, Newman AR, Slutsman J, Hinds PS. Surprised by Benefit in Pediatric Palliative Care Research. Cancer Nurs. 2018 Jan/Feb;41(1):86-87. doi: 10.1097/NCC.0000000000000576. No abstract available. PMID 29206683
- [Background] Needle JS, Peden-McAlpine C, Liaschenko J, Koschmann K, Sanders N, Smith A, Schellinger SE, Lyon ME. "Can you tell me why you made that choice?": A qualitative study of the influences on treatment decisions in advance care planning among adolescents and young adults undergoing bone marrow transplant. Palliat Med. 2020 Mar;34(3):281-290. doi: 10.1177/0269216319883977. Epub 2019 Oct 29. PMID 31659933
- [Background] Wiener L, Zadeh BS, Battles H, Sender L, Fasciano K, Heath C, Lyon ME, Donavan KA, Naronoha Ferrazde Arruda Colli M, Pao M. Courageous Conversations: Advance Care Planning and Family Communication. Pediatric Blood & Cancer, S596, October, 2018
- [Result] Curtin KB, Watson AE, Wang J, Okonkwo OC, Lyon ME. Pediatric advance care planning (pACP) for teens with cancer and their families: Design of a dyadic, longitudinal RCCT. Contemp Clin Trials. 2017 Nov;62:121-129. doi: 10.1016/j.cct.2017.08.016. Epub 2017 Aug 24. PMID 28844985
- [Result] Gaines ThompkinsJ, Friebert S, Baker J, Needle J, Cheng Y, Lyon M. Effect of FAmily CEntered (FACE) advance care planning (ACP) on families' appraisals of caregiving for their teens with cancer. J Pain Symptom Manage 2019;57(2):446-447. PMID: 30267845
- [Result] Friebert S, Gaines (Thompkins) J, Needle J, Baker J, Cheng Y, Lyon M. What do adolescents want? Values, goals and beliefs of teens with cancer. J Pain Symptom Manage 2019;57(2):378.
- [Result] Grossoehme DH, Friebert S, Baker JN, Tweddle M, Needle J, Chrastek J, Thompkins J, Wang J, Cheng YI, Lyon ME. Association of Religious and Spiritual Factors With Patient-Reported Outcomes of Anxiety, Depressive Symptoms, Fatigue, and Pain Interference Among Adolescents and Young Adults With Cancer. JAMA Netw Open. 2020 Jun 1;3(6):e206696. doi: 10.1001/jamanetworkopen.2020.6696. PMID 32543698
- [Result] Friebert S, Grossoehme DH, Baker JN, Needle J, Thompkins JD, Cheng YI, Wang J, Lyon ME. Congruence Gaps Between Adolescents With Cancer and Their Families Regarding Values, Goals, and Beliefs About End-of-Life Care. JAMA Netw Open. 2020 May 1;3(5):e205424. doi: 10.1001/jamanetworkopen.2020.5424. PMID 32427325
- [Result] Thompkins J, Baker JN, Friebert S, Needle J, Wang J, Cheng YI, Lyon ME. Effect of FAmily CEnterd (FACE) advance care planning (ACP) on families' appraisals of caregiving for their teen with cancer. 2020 American Society of Clinical Oncology (ASCO) Annual Meeting. (ASCO Virtual Scientific Program). J Clin Oncol 38: 2020 (suppl; abstr e22533) DOI:10.1200/JCO.2020.38.15_suppl.e2253
- [Result] Schreiner K, Grossoehme DH, Friebert S, Baker JN, Needle J, Lyon ME. "Living life as if I never had cancer": A study of the meaning of living well in adolescents and young adults who have experienced cancer. Pediatr Blood Cancer. 2020 Oct;67(10):e28599. doi: 10.1002/pbc.28599. Epub 2020 Jul 19. PMID 32686240
- [Result] Livingston J, Cheng Y, Wang J, Tweddle T, Friebert S, Baker J, Thompkins J, Greenberg I, Lyon M. FP029 SIOP19-1654 Shared Spiritual Beliefs Between Adolescents with Cancer and Their Families: An Exploration of Social Determinants of Spiritual Well-Being. Supplement: Abstracts from the 51st Congress of the International Society of Paediatric Oncology (SIOP) Lyon, France, October 23-26, 2019 Pediatric Blood & Cancer. December 2019;66: IssueS4 e27989 https://doi.org/10.1002/pbc.27989
- [Result] Thompkins J, Greenberg I, Cheng Y, Baker J, Needle J, Friebert S, Tweddle M, Wang J, Lyon M. FP030 SIOP19-1630 The Influence of Religious Beliefs on Symptoms of Anxiety and Depression Among Adolescents with Cancer Supplement: Abstracts from the 51st Congress of the International Society of Paediatric Oncology (SIOP) Lyon, France, October 23-26, 2019 Pediatric Blood & Cancer. December 2019;66: IssueS4 e27989 https://doi.org/10.1002/pbc.27989
- [Result] Lyon ME, Grossoehme DH, Baker JN, Friebert S, Cheng Y, Chrastek J, Thompkins J, Tweddle M, Wang J, Needle J. Relationship of spiritual constructs to mental health PROs in adolescents with cancer.DOI: 10.1200/JCO.2019.37.31_suppl.136 Journal of Clinical Oncology 37, no. 31_suppl (November 01, 2019) 136-136. Published online November 25, 2019
- [Result] Needle JS, Friebert S, Thompkins JD, Grossoehme DH, Baker JN, Jiang J, Wang J, Lyon ME. Effect of the Family-Centered Advance Care Planning for Teens with Cancer Intervention on Sustainability of Congruence About End-of-Life Treatment Preferences: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2220696. doi: 10.1001/jamanetworkopen.2022.20696. PMID 35819787
- [Result] Baker JN, Friebert S, Needle J, Jiang J, Wang J, Lyon ME. An Intervention in Congruence for End-of-Life Treatment Preference: A Randomized Trial. Pediatrics. 2022 May 1;149(5):e2021054796. doi: 10.1542/peds.2021-054796. PMID 35425986
- [Result] Thompkins JD, Needle J, Baker JN, Briggs L, Cheng YI, Wang J, Friebert S, Lyon ME. Pediatric Advance Care Planning and Families' Positive Caregiving Appraisals: An RCT. Pediatrics. 2021 Jun;147(6):e2020029330. doi: 10.1542/peds.2020-029330. Epub 2021 May 6. PMID 33958436
- [Result] - Baker JN (presenter), Friebert S, Needle JS, Thompkins JD, Grossoehme D, Jiang J, Wang J, Lyon ME. Oral Presentation. The effect of Family-Centered pediatric Advance Care Planning for Teens with Cancer (FACE®-TC) on adolescents' decisional support, preparedness, and symptoms at 3- and 12- months post-intervention. 54th Congress of the International Society of Paediatric Oncologists (SIOP). September 29, 2022. Barcelona, Spain
- [Result] Lyon ME, Cheng YI, Needle J, Friebert S, Baker JN, Jiang J, Wang J. The intersectionality of gender and poverty on symptom suffering among adolescents with cancer. Pediatr Blood Cancer. 2021 Aug;68(8):e29144. doi: 10.1002/pbc.29144. Epub 2021 Jun 1. PMID 34061435
- [Result] Livingston J, Cheng YI, Wang J, Tweddle M, Friebert S, Baker JN, Thompkins J, Lyon ME. Shared spiritual beliefs between adolescents with cancer and their families. Pediatr Blood Cancer. 2020 Dec;67(12):e28696. doi: 10.1002/pbc.28696. Epub 2020 Sep 12. PMID 32918519
- [Result] Friebert S, Trujillo Rivera EA, Baker JN, Thompkins JD, Grossoehme D, Needle J, Lyon ME. Pediatric Advance Care Planning and Adolescent Preparedness and Quality of Life: An RCT. Pediatrics. 2025 Feb 1;155(2):e2024068699. doi: 10.1542/peds.2024-068699. PMID 39821687

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 260 participants enrolled in the study. Randomization was at the level of the dyad (adolescent with cancer and family surrogate decision maker). After enrollment a secondary screening occurred. 4 participants who were part of an adolescent/family dyad (n=8 participants) failed this secondary screening. Thus, 252 participants (126 adolescent/family dyads) completed the baseline assessment and were then randomized. The flow chart is reported as adolescent/family dyads.
Period: Overall Study
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Started (2:1 ratio FACE-TC to TAU) | 83 (numbers reflect adolescent/family dyads) | 43 (numbers reflect adolescent/family dyads)
Completed | 66 (numbers reflect adolescent/family dyads) | 38 (numbers reflect adolescent/family dyads)
Not Completed | 17 | 5
Not completed — Death | 3 | 2
Not completed — Lost to Follow-up | 7 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — patient wanted to leave it behind | 1 | 0
Not completed — anxiety | 1 | 0
Not completed — family issues | 1 | 0
Not completed — no reason given | 1 | 0

BASELINE CHARACTERISTICS:
Population: 260 participants were consented/assented and enrolled. Upon secondary screening 8 participants were excluded, leaving 252 participants. Participants were randomized as adolescent/family surrogate dyads at 2:1 ratio of intervention (n=83 dyads) to control (n=43 dyads). Baseline analysis was at level of participant with separate analysis for adolescents and family surrogates. Outcome measure for Statement of Treatment Preferences (SOTP) was at level of the dyad and not administered at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU) | Total
Number analyzed (Participants) | 166 | 86 | 252
Age, Categorical [Count of Participants; unit: Participants] — Population: Row population represents analysis by adolescents separately from family surrogate decision makers. Secondary analysis was conducted with each group separately. Primary outcome was congruence in treatment preferences and analysis was at the level of the adolescent/family dyad.
  Participants
    adolescents: number analyzed (Participants) | 83 | 43 | 126
    adolescents: <=18 years | 44 | 25 | 69
    adolescents: Between 18 and 65 years | 39 | 18 | 57
    adolescents: >=65 years | 0 | 0 | 0
    family surrogates: number analyzed (Participants) | 83 | 43 | 126
    family surrogates: <=18 years | 0 | 0 | 0
    family surrogates: Between 18 and 65 years | 81 | 43 | 124
    family surrogates: >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years]
  Adolescents | 16.9 [14 to 20] | 17.0 [14 to 20] | 17 [14 to 20]
  Family surrogate | 45.6 [19 to 67] | 46.5 [20 to 63] | 46 [19 to 67]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex is by self-report. Population: Age of adolescents and family surrogate decision makers were used as separate variables in the analysis.
  Participants
    adolescents: number analyzed (Participants) | 83 | 43 | 126
    adolescents: Female | 45 | 27 | 72
    adolescents: Male | 38 | 16 | 54
    family surrogates: number analyzed (Participants) | 83 | 43 | 126
    family surrogates: Female | 67 | 37 | 104
    family surrogates: Male | 16 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was analyzed as a separate variable for adolescents and family surrogates.
  Participants
    adolescents: number analyzed (Participants) | 83 | 43 | 126
    adolescents: Hispanic or Latino | 5 | 0 | 5
    adolescents: Not Hispanic or Latino | 76 | 40 | 116
    adolescents: Unknown or Not Reported | 2 | 3 | 5
    family surrogates: number analyzed (Participants) | 83 | 43 | 126
    family surrogates: Hispanic or Latino | 4 | 0 | 4
    family surrogates: Not Hispanic or Latino | 79 | 42 | 121
    family surrogates: Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was measured by self-report. Population: Race of adolescents did not always match race of family surrogate. Therefore, the variables were analyzed separately.
  Participants
    adolescents: number analyzed (Participants) | 83 | 43 | 126
    adolescents: American Indian or Alaska Native | 0 | 0 | 0
    adolescents: Asian | 3 | 0 | 3
    adolescents: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    adolescents: Black or African American | 12 | 5 | 17
    adolescents: White | 63 | 37 | 100
    adolescents: More than one race | 4 | 1 | 5
    adolescents: Unknown or Not Reported | 1 | 0 | 1
    family surrogates: number analyzed (Participants) | 83 | 43 | 126
    family surrogates: American Indian or Alaska Native | 0 | 1 | 1
    family surrogates: Asian | 3 | 0 | 3
    family surrogates: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    family surrogates: Black or African American | 10 | 4 | 14
    family surrogates: White | 68 | 35 | 103
    family surrogates: More than one race | 2 | 3 | 5
    family surrogates: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 166 | 86 | 252
Patient-Reported Outcomes Measures Short Forms pediatric [Median (Inter-Quartile Range); unit: units on a scale] — pediatric PROMIS Short Forms 8a - Pediatrics v. 2.0) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in children and adolescents. Assessed adolescent Emotional distress-Anxiety; Emotional Distress-Depressive Symptoms; Fatigue; and Pain Interference using these PROMIS subscales. Each subscale has 8 items each. Minimum value is 8. Maximum value is 40. Higher scores mean worse outcomes for anxiety, depressive symptoms, fatigue, and pain interference. Measures were administered to adolescents only. Population: Adolescents living with cancer only. There are no missing data. The numbers analyzed in some rows differ from the Overall Number of Participants Analyzed for this Outcome Measure due either to missed study visits or attrition.
  units on a scale
    Emotional Distress - Anxiety: number analyzed (Participants) | 83 | 43 | 126
    Emotional Distress - Anxiety | 13.0 [10 to 16.5] | 12.0 [9.0 to 18.0] | 13.0 [10.0 to 17.8]
    Emotional Distress - Depressive Symptoms: number analyzed (Participants) | 83 | 43 | 126
    Emotional Distress - Depressive Symptoms | 10.0 [8.0 to 16.0] | 10.0 [8.0 to 13.5] | 10.0 [8.0 to 15.8]
    Fatigue: number analyzed (Participants) | 83 | 43 | 126
    Fatigue | 16.0 [11.0 to 23.0] | 15.0 [12.0 to 22.5] | 16.0 [11.0 to 23.0]
    Pain Interference: number analyzed (Participants) | 83 | 43 | 126
    Pain Interference | 10.0 [8.0 to 16.0] | 10.0 [8.0 to 20.5] | 10.0 [8.0 to 17.0]
Family Appraisal of Caregiving Questionnaire for Palliative Care [Mean (Standard Deviation); unit: units on a scale] — FACQ-PC is a 25-item measure consisting of four subscales:(i) caregiver strain, (ii) positive caregiving appraisals, (iii) caregiver distress, and (iv) family well-being. Scores are from 5 = strongly agree to 1 = strongly disagree. We did not calculate a Total score. The FACQ-PC subscale scores were computed by taking the mean of the items (score range 1-5). Some items were reverse scored, depending on how the item is phrased, so that higher scores = higher amount of the subscale being measured. Minimum value for each subscale is 1 and the maximum value for each subscale is 5. Population: Row population differs from overall, because only family member completed this questionnaire and because of attrition from time of enrollment.
  units on a scale
    Caregiver strain: number analyzed (Participants) | 83 | 43 | 126
    Caregiver strain | 2.17 (0.75) | 2.34 (0.89) | 2.23 (0.80)
    Positive Caregiving Appraisal: number analyzed (Participants) | 83 | 43 | 126
    Positive Caregiving Appraisal | 4.51 (0.46) | 4.61 (0.40) | 4.54 (0.44)
    Caregiver distress: number analyzed (Participants) | 83 | 43 | 126
    Caregiver distress | 2.19 (0.78) | 2.44 (0.80) | 2.28 (0.79)
    Family well-being: number analyzed (Participants) | 83 | 43 | 126
    Family well-being | 4.13 (0.67) | 4.25 (0.63) | 4.17 (0.66)
Functional Assessment of Chronic Illness Therapy (FACIT)-Spirituality-12 Version 4 Expanded [Median (Inter-Quartile Range); unit: units on a scale] — Assessed spiritual well-being. Subscales Meaning/Peace (7 items) and Faith (5 items) and Total score (12 items) were calculated on a 5-point Likert scale from 0=not at all to 5=very much. Some items are reverse scored. See www.facit.org Meaning/Peace subscale score range from minimum value of 0 to maximum value of 32. Higher scores indicate better meaning/peace. Faith subscale score range from 0 minimum value to maximum value of 16. Higher scores indicate greater faith. Total score range is from 0 minimum value to maximum value of 92. Higher scores indicate better spiritual well-being. Population: Scores are reported separately for adolescents and the family member. Total participants completing FACIT-SP is 252. The other discrepancy is caused by attrition between enrollment and baseline visit.
  units on a scale
    Adolescent Meaning/Peace: number analyzed (Participants) | 83 | 43 | 126
    Adolescent Meaning/Peace | 28.0 [25.0 to 30.0] | 26.0 [23.5 to 29.0] | 28.0 [24.0 to 30.0]
    Adolescent Faith: number analyzed (Participants) | 83 | 43 | 126
    Adolescent Faith | 12.0 [9.0 to 15.5] | 14.0 [9.0 to 15.5] | 12.5 [9.0 to 15.8]
    Adolescent Total score: number analyzed (Participants) | 83 | 43 | 126
    Adolescent Total score | 78.0 [69.5 to 85.5] | 75.0 [69.0 to 82.0] | 77.0 [69.3 to 85.0]
    Family Meaning/Peace: number analyzed (Participants) | 83 | 43 | 126
    Family Meaning/Peace | 28.0 [26.0 to 30.0] | 29.0 [27.0 to 32.0] | 28.0 [26.0 to 30.0]
    Family Faith: number analyzed (Participants) | 83 | 43 | 126
    Family Faith | 13.0 [10.0 to 16.0] | 15.0 [12.0 to 16.0] | 14.0 [11.0 to 16.0]
    Family Total score: number analyzed (Participants) | 83 | 43 | 126
    Family Total score | 79.0 [71.5 to 84.5] | 85.0 [75.5 to 89.0] | 80.5 [72.3 to 87.0]

OUTCOME MEASURES:

1. Primary Outcome: Statement of Treatment Preferences (SOTP) a Tool to Measure Goals of Care.
Description: Statement of Treatment Preferences documented adolescents' goals of care and families' understanding. Situations were: (1) prolonged hospital stay with ongoing medical intervention and low chance of survival; (2) treatments extend life by no more than 2-3 months with side-effects; (3) physical impairment; and (4) mental impairment. Choices for the four situations were "to continue all treatments …", "to stop all efforts to keep me alive…", or "do not know." Responses for data analysis were recoded into two categories: congruent (family accurately reported what the patient reported as their treatment preference) versus "stop all treatments." Dyadic responses, "do not know" were treated as not congruent and removed from analysis. Percentage dyadic agreement or disagreement was calculated for each situation. Minimum agreement is 0%. Maximum agreement is 100%. Higher percentage dyadic agreement is better outcome.
Time Frame: Agreement on SOTP was assessed 2 weeks post-baseline for controls or immediately following Session 2 for FACE-TC intervention dyads, and at 3, 6, 12 and 18 months.
Population: Total number for overall congruence of Statement of Treatment Preferences 2-weeks post baseline or post-Session 2 (n=115 dyads). Data were analyzed and are presented at the level of dyadic congruence, i.e. 73 dyads (146 adolescent and family participants) in the intervention arm and 42 dyads (84 participants) in the control arm. 1 dyad (2 participants) had missing data.
Measure: Count of Units; unit: Dyads
Units Other Than Participants: Dyads
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 146 | 84
Number analyzed (Dyads) | 73 | 42
Dyads
  Immediately post-session 2: Poor Agreement: Agree 0-1 situation | 10 | 22
  Immediately post-session 2: Moderate Agreement: Agree 2-3 situations | 38 | 19
  Immediately post-session 2: Perfect agreement: agree all 4 situations | 25 | 1
  3 Months post-intervention: number analyzed (Participants) | 130 | 74
  3 Months post-intervention: number analyzed (Dyads) | 65 | 37
  3 Months post-intervention: Poor Agreement: Agree 0-1 situation | 23 | 12
  3 Months post-intervention: Moderate Agreement: Agree 2-3 situations | 37 | 19
  3 Months post-intervention: Perfect agreement: agree all 4 situations | 5 | 6
Statistical Analysis 1: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Analysis was at the level of the dyad. AIM 1. To evaluate the efficacy of FACE-TC on patient-family congruence in treatment preferences. H1a: FACE-TC participants will better maintain congruence over time, compared to controls. H1b: Development of congruence may not be homogeneous and FACE-TC may influence the pattern of congruence development; Test type: Superiority — First measure of congruence was taken at 2 weeks post-baseline for controls, or immediately post-Session 2 for intervention dyads. Analysis presented here assessed differences between groups in agreement. This represents the underlying data without examining the pattern of congruence for each dyad over time. Longitudinal latent class analysis of congruence in responses over time between adolescents/families was conducted at the person not variable level; p < 0.05, longitudinal latent class analysis; examined the pattern of change over time; Odds Ratio (OR) = 3.22, 95% CI 2-sided [1.09 to 9.57]

2. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS Short Forms 8a - Pediatrics v. 2.0) is a Set of Person-centered Measures That Evaluates and Monitors Physical, Mental, and Social Health in Children and Adolescents.
Description: Assessed adolescent Emotional distress-Anxiety; Emotional Distress-Depressive Symptoms; Fatigue; and Pain Interference using these PROMIS subscales. Each subscale has 8 items each. Minimum value is 8. Maximum value is 40. Higher scores mean worse outcomes for anxiety, depressive symptoms, fatigue, and pain interference.
Time Frame: Change from baseline in quality of life (defined as symptoms of anxiety, depression, fatigue and pain interference) at 3, 6, and 12 months post baseline compared to controls
Population: Adolescents living with cancer. Higher scores indicate worse symptoms of anxiety, depressive symptoms, fatigue and pain interference. There are no missing data. The numbers analyzed in some rows differ from the Overall Number of Participants Analyzed for this Outcome Measure due either to missed study visits, attrition, or deaths at 3-months, 6-months, and 12-months. Changes in number of participants reflects missing visits, deaths, or attrition.
Measure: Median (Inter-Quartile Range); unit: raw score units on a scale
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 83 | 43
raw score units on a scale
  Emotional Distress-Anxiety baseline | 13.0 [10.0 to 16.5] | 12.0 [9.0 to 18.0]
  Emotional Distress -Depressive Symptoms symptoms baseline | 10.0 [8.0 to 16.0] | 10.0 [8.0 to 13.5]
  Fatigue baseline | 16.0 [11.0 to 23.0] | 15.0 [12.0 to 22.5]
  Pain Interference baseline | 10.0 [8.0 to 16.0] | 10.0 [8.0 to 20.5]
  Emotional Distress Anxiety 3 months: number analyzed (Participants) | 67 | 40
  Emotional Distress Anxiety 3 months | 17 [12 to 22] | 12.5 [10.0 to 20.0]
  Emotional Distress Depressive Symptoms 3 Months: number analyzed (Participants) | 67 | 40
  Emotional Distress Depressive Symptoms 3 Months | 13.0 [8.0 to 21.0] | 11.0 [8.0 to 18.5]
  Fatigue 3 months: number analyzed (Participants) | 67 | 40
  Fatigue 3 months | 18 [12.0 to 31.0] | 14.0 [10.0 to 21.0]
  Pain Interference 3 months: number analyzed (Participants) | 67 | 40
  Pain Interference 3 months | 12.0 [8.0 to 21.0] | 10.5 [8.0 to 16.0]
  Emotional distress - anxiety 6 months: number analyzed (Participants) | 67 | 41
  Emotional distress - anxiety 6 months | 16.0 [12.0 to 21.0] | 14.0 [11.0 to 21.0]
  Emotional distress - depressive symptoms 6 months: number analyzed (Participants) | 67 | 41
  Emotional distress - depressive symptoms 6 months | 13.0 [8.0 to 19.0] | 10.0 [8.0 to 15.0]
  Fatigue 6 months: number analyzed (Participants) | 67 | 41
  Fatigue 6 months | 16.0 [11.0 to 29.0] | 16.0 [11.0 to 25.0]
  Pain Interference 6 months: number analyzed (Participants) | 67 | 41
  Pain Interference 6 months | 11.0 [8.0 to 19.0] | 9.0 [8.0 to 15.0]
  Emotional distress - anxiety 12 months: number analyzed (Participants) | 66 | 38
  Emotional distress - anxiety 12 months | 17.0 [11.0 to 22.0] | 11.0 [8.8 to 18.0]
  Emotional distress - depression: number analyzed (Participants) | 66 | 38
  Emotional distress - depression | 12.0 [9.0 to 19.3] | 10.0 [8.0 to 13.3]
  Fatigue - 12 months: number analyzed (Participants) | 66 | 38
  Fatigue - 12 months | 17.0 [10.0 to 27.0] | 12.5 [10.0 to 21.3]
  Pain Interference - 12 months: number analyzed (Participants) | 66 | 38
  Pain Interference - 12 months | 10.5 [8.0 to 18.0] | 8.0 [8.0 to 12.0]
Statistical Analysis 1: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Emotional distress-anxiety analysis at baseline comparing intervention and control; Test type: Superiority; p < 0.05, Mixed Models Analysis — The generalized mixed effect models are taking into account missingness by attrition. There were not missing values for the outcomes or predictors that we used; Model forced age, gender, race, family education, family income under the Federal Poverty level, on/off treatment; Risk Ratio (RR) = 1.00743162, 95% CI 2-sided [0.928 to 1.094]
Statistical Analysis 2: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Emotional distress-anxiety analysis at 3 months post baseline comparing intervention and control. We hypothesized that anxiety would be lower in the intervention group compared to controls; Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Model forced age, gender, race, family education, family income under the Federal Poverty level, on/off treatment; Risk Ratio (RR) = 1.05037501, 95% CI 2-sided [0.96438584 to 1.14403138]
Statistical Analysis 3: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); This is analysis for 6 month outcomes of Emotional-distress - anxiety. See details in 3 month outcomes; Test type: Superiority — See earlier comments; p < 0.05, t-test, 2 sided — See earlier comments; See earlier comments; Risk Ratio (RR) = 1.01136067, 95% CI 2-sided [0.92887892 to 1.10116656]
Statistical Analysis 4: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); These are the 12 month outcomes for Emotional distress - anxiety. See earlier comments; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 1.14070431, 95% CI 2-sided [1.04444724 to 1.24583250] — See earlier comments
Statistical Analysis 5: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); This analysis is for the outcome Emotional distress - depressive symptoms. We hypothesized that adolescent in the intervention would have lower depressive symptoms compared to controls at 3, 6, and 12 month outcomes. The following are the baseline comparisons between control and intervention which were controlled for in the 3, 6, and 12 month analysis of outcomes; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 0.98078271, 95% CI 2-sided [0.89845609 to 1.07065301]
Statistical Analysis 6: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); The results here are for the outcome variable Emotional Distress - Depressive symptoms at 3 month outcomes. We hypothesized that adolescents randomized to the intervention would have lower depressive symptoms than controls; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 1.04007715, 95% CI 2-sided [0.94970156 to 1.13905306]
Statistical Analysis 7: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); We hypothesize that Emotional Distress - Depressive symptoms would be lower in intervention adolescents compared to controls at 6 months post intervention; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 1.07347088, 95% CI 2-sided [0.98062710 to 1.17510491]
Statistical Analysis 8: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); We hypothesized that adolescents randomized to the intervention would have lower scores on Emotional Distress - Depressive symptoms compared to controls at 12 months post baseline; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 1.11582434, 95% CI 2-sided [1.01653156 to 1.22481585]
Statistical Analysis 9: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); We hypothesized that adolescents randomized to the intervention would have no differences in fatigue at baseline if randomization was successful. In this analysis we examine the baseline results; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio, log = 0.98803061, 95% CI 2-sided [0.89065531 to 1.09605195]
Statistical Analysis 10: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); We hypothesized that adolescents randomized to the intervention arm would report less Fatigue at 3 months outcome compared to controls; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 1.13509797, 95% CI 2-sided [1.01959639 to 1.26368376]
Statistical Analysis 11: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); We hypothesized that adolescents randomized to the intervention would report less Fatigue at 6 months post baseline compared to control adolescents; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 1.04944737, 95% CI 2-sided [0.94281417 to 1.16814089]
Statistical Analysis 12: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); We hypothesized that intervention adolescents would report less Fatigue than controls at 12 months post baseline; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 1.11042568, 95% CI 2-sided [0.99383841 to 1.24068981]
Statistical Analysis 13: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); We hypothesized that there would be no differences at baseline between intervention and control adolescents with respect to Pain Interference; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 0.96833470, 95% CI 2-sided [0.88658183 to 1.05762611]
Statistical Analysis 14: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); We hypothesized that adolescents randomized to the intervention compared to controls would report less Pain Interference at 3 months post baseline; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 1.04450374, 95% CI 2-sided [0.95307464 to 1.14470370]
Statistical Analysis 15: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); We hypothesized that adolescents randomized to the intervention compared to controls would report less Pain Interference at 6 months post baseline; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 1.07182133, 95% CI 2-sided [0.97835451 to 1.17421748]
Statistical Analysis 16: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); We hypothesized that at 12 month outcome adolescents randomized to the intervention would report less Pain Interference compared to control adolescents; Test type: Superiority; p < 0.05, t-test, 2 sided; Risk Ratio, log = 1.09964781, 95% CI 2-sided [1.00051223 to 1.20860622]

3. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Spirituality-12 Version 4 Expanded (FACIT-Sp-EX)
Description: Assessed construct of spiritual well-being. Two subscales Meaning/Peace (7 items) and Faith (5 items) and Total score (12 items) were calculated. on a 5-point Likert scale from 0=not at all to 5=very much. Some items are reverse scored. See www.facit.org Meaning/Peace subscale score range from minimum value of 0 to maximum value of 32. Higher scores indicate better meaning/peace.
  Faith subscale score range from 0 minimum value to maximum value of 16. Higher scores indicate better meaning/peace.
  Total score range is from 0 minimum value to maximum value of 92. Higher scores indicate better spiritual well-being.
Time Frame: Controlling for baseline, change in of meaning and peace subscale and faith subscale at 3, 6, 12 months post intervention for intervention adolescents compared to control adolescents. Total scores provided for interested investigators were not outcome.
Population: Adolescents living with cancer. The numbers analyzed in some rows differ from the Overall Number of Participants Analyzed for this Outcome Measure due to missed study visits, attrition, or deaths at 3-months, 6-months, and 12-months. There are no missing data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 83 | 43
units on a scale
  Meaning and Peace subscale baseline | 28.0 [25.0 to 30.0] | 26.0 [23.5 to 29.0]
  Faith subscale baseline | 12.0 [9.0 to 15.5] | 14.0 [9.0 to 15.5]
  Total FACIT-SP vs. 4 score baseline | 78 [69.5 to 85.5] | 75.0 [69.0 to 82.0]
  Meaning and Peace subscale 3 months: number analyzed (Participants) | 67 | 40
  Meaning and Peace subscale 3 months | 26.0 [23.0 to 30.0] | 27.5 [22.3 to 29.0]
  Faith subscale 3 months: number analyzed (Participants) | 67 | 40
  Faith subscale 3 months | 12.0 [8.0 to 15.0] | 12.0 [9.3 to 15.0]
  FACIT-SP vs4 Total Score 3 months: number analyzed (Participants) | 67 | 40
  FACIT-SP vs4 Total Score 3 months | 72.0 [65.0 to 84.0] | 75.0 [66.0 to 86.0]
  Meaning and Peace subscale 6 months: number analyzed (Participants) | 67 | 41
  Meaning and Peace subscale 6 months | 26.0 [24.0 to 30.0] | 27.0 [24.0 to 31.0]
  Faith subscale 6 months: number analyzed (Participants) | 67 | 41
  Faith subscale 6 months | 12.0 [6.0 to 15.0] | 12.0 [7.0 to 15.0]
  FACIT-Sp v4 Total score 6 months: number analyzed (Participants) | 67 | 41
  FACIT-Sp v4 Total score 6 months | 76.0 [64.0 to 83.0] | 77.0 [61.0 to 84.0]
  Meaning and Peace subscale 12 month: number analyzed (Participants) | 66 | 38
  Meaning and Peace subscale 12 month | 26.0 [23.0 to 30.0] | 29.5 [25.0 to 32.0]
  Faith subscale 12 months: number analyzed (Participants) | 66 | 38
  Faith subscale 12 months | 11.0 [8.0 to 16.0] | 12.0 [8.0 to 16.0]
  FACIT-SP v4 Total 12 months: number analyzed (Participants) | 66 | 38
  FACIT-SP v4 Total 12 months | 71 [62.0 to 82.0] | 80.5 [68.8 to 88.0]
Statistical Analysis 1: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Meaning and Peace Subscale at 3 months post intervention; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean ratio = 0.98, 95% CI 2-sided [0.88 to 1.09]
Statistical Analysis 2: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Meaning and Peace subscale at 6 months post intervention; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean ratio = 0.97, 95% CI 2-sided [0.88 to 1.08]
Statistical Analysis 3: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Meaning and Peace subscale at 12 months post intervention; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean ratio = 0.92, 95% CI 2-sided [0.82 to 1.02]
Statistical Analysis 4: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Faith subscale score at 3 months post intervention; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean ratio = 0.92, 95% CI 2-sided [0.73 to 1.16]
Statistical Analysis 5: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Faith subscale at 6 months post intervention; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean ratio = 0.96, 95% CI 2-sided [0.76 to 1.21]
Statistical Analysis 6: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Faith subscale scores at 12 months post intervention; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean ratio = 0.92, 95% CI 2-sided [0.72 to 1.17]

4. Secondary Outcome: Family Appraisal of Caregiving Questionnaire for Palliative Care (FACQ-PC)
Description: The FACQ-PC is a 25-item measure consists of four theoretically derived subscales: (i) caregiver strain, (ii) positive caregiving appraisals, (iii) caregiver distress, and (iv) family well-being. Scores are from 5 = strongly agree to 1 = strongly disagree. We did not calculate a Total score. We only used the 4 subscale scores. On the subscale scores for positive caregiving appraisals and family well-being, higher scores mean better outcomes, i.e. greater positive caregiving appraisals or family well-being. On the subscale scores for caregiver strain and caregiver distress, higher scores mean worse outcomes, i.e. greater caregiver strain or caregiver distress. The FACQ-PC subscale scores were computed by taking the mean of the items (score range 1-5). Some items were reverse scored, depending on how the item is phrased, so that higher scores = higher amount of the subscale being measured. So the minimum value for each subscale is 1 and the maximum value for each subscale is 5.
Time Frame: Baseline and 3 months post baseline administered to family surrogates only.
Population: Data were analyzed for family surrogate only. 83 surrogates randomized to FACE TC and 43 surrogates randomized to TAU at baseline. At 3 months post-intervention analyzed population was 65 FACE-TC and 37 TAU. One TAU surrogate missed this study visit at 3 months post intervention. Changes in number of participants reflect missed study visits, deaths, or loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 83 | 43
units on a scale
  Caregiver strain Baseline | 2.17 (0.75) | 2.34 (0.89)
  Positive Caregiving Appraisal Baseline | 4.51 (0.46) | 4.61 (0.40)
  Caregiver distress Baseline | 2.19 (0.78) | 2.44 (0.80)
  Family Wellbeing (Higher score=better wellbeing) | 4.13 (0.67) | 4.25 (0.63)
  Caregiver strain 3 months | 2.15 (0.81) | 2.39 (0.81)
  Positive caregiving appraisal 3 months | 4.55 (0.45) | 4.47 (0.54)
  Caregiver distress 3 months | 2.23 (0.90) | 2.49 (1.01)
  Family well-being 3 months | 4.12 (0.70) | 4.09 (0.67)
Statistical Analysis 1: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Caregiver Strain subscale at 3 months post-intervention comparing intervention to TAU, controlling for baseline levels; Test type: Superiority; p < 0.05, GEE model; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.42 to 0.15]
Statistical Analysis 2: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Positive Caregiving Appraisal subscale at 3 months post-intervention comparing intervention to TAU, controlling for baseline levels; Test type: Superiority; p < 0.05, GEE model; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.02 to 0.36]
Statistical Analysis 3: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Caregiver Distress subscale at 3 months post-intervention comparing intervention to TAU, controlling for baseline levels; Test type: Superiority; p < 0.05, GEE model; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.35 to 0.32]
Statistical Analysis 4: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Family Well-Being subscale at 3 months post-intervention, comparing intervention to TAU, controlling for baseline levels; Test type: Superiority; p < 0.05, GEE model; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.07 to 0.38]

5. Secondary Outcome: Advance Directive for Adolescent Only Located in the Electronic Health Record at Study Close Out.
Description: The effect of the intervention on documentation in the Electronic Health Record of any advance directive for the adolescent was conducted at study close, using a standardized chart abstraction form.
Time Frame: This adolescent outcome was measured at one time point only, between 18 months post-intervention or study close-out. At study close out we had 117 adolescents in the study. Attrition was due to deaths, lost to follow-up, and withdrawals.
Population: Adolescent data only on documentation of an advance directive in the electronic health.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 75 | 42
Participants
  Any advance directive, yes | 60 | 8
  Any advance directive, no | 15 | 34

6. Other Pre Specified Outcome: Quality of End of Life Communication (QOC)
Description: Curtis's Quality of Participant-Interviewer Communication Questionnaire (Curtis et al 1999) evaluated quality of communication that occurred between participants and facilitator. The first 4 items are: 1. Do you think that your attitudes are known by the interviewer? 2. Did you feel that the interviewer cared about you as a person? 3. Did you feel that the interviewer listened to what you said? 4. Did you feel that the interviewer gave you enough attention? 5-point Likert scale ranging from Probably no to probably yes.
  The 5th item is: How would you rate the overall quality of the discussions you just had with the interviewer? Range of scores is from 5 to 25. Higher scores indicate higher quality of communication.
Time Frame: 234 participants completed this assessment at two weeks post-baseline for control; two weeks post-baseline for intervention--immediately following Session 2. This process assessment is not in the flow diagram because it is not an intervention outcome.
Population: Participants (adolescents with cancer and their family surrogate decision-maker) ratings of quality of communication with facilitator. Separate analysis were conducted for adolescents and their family surrogate, i.e. analysis was not at the level of the dyad. Changes in participants over time reflect missed study visits, deaths, or loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 150 | 84
units on a scale
  Adolescent ratings: number analyzed (Participants) | 75 | 42
  Adolescent ratings | 22.3 (3.2) | 22.1 (2.4)
  Family member ratings: number analyzed (Participants) | 75 | 42
  Family member ratings | 23.4 (1.8) | 22.4 (2.4)
Statistical Analysis 1: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Quality of communication analysis for adolescents; Test type: Superiority; p = 0.47, Regression, Linear; Intervention effect for quality of adolescent communication score controlling for age, gender, race, income and on active treatment; Slope = 0.44, Standard Error of Mean 0.59 — It is the standard error of the slope, but this was not an option
Statistical Analysis 2: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Quality of communication analysis for family member; Test type: Superiority; p < 0.01, Regression, Linear; Testing intervention effect for family member quality of communication score controlling for age, gender, race, income nd on active treatment; Slope = 1.15, Standard Error of Mean 0.41 — This is standard error of the slope

7. Other Pre Specified Outcome: Brief Multidimensional Measurement of Religiousness/Spirituality (BMMRS-adapted)
Description: Responses to "How often do you go to religious services? Responses ranged from "more than once a week" to "once or twice a year." Higher scores indicated greater attendance at religious services. Responses were used as a covariate in the initial Generalized linear mixed effect models. Prior research had indicated that this variable moderated quality of life outcomes.
Time Frame: Assessed at baseline and at 3, 6, and 12 months post-intervention.
Population: Adolescents with cancer responses at baseline, 3, 6 and 12 months post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 83 | 43
Participants
  Baseline: Declined | 2 | 1
  Baseline: Every month or so | 6 | 5
  Baseline: Every week or more often | 20 | 10
  Baseline: More than once a week | 8 | 3
  Baseline: Never | 13 | 9
  Baseline: Once or twice a month | 21 | 9
  Baseline: Once or twice a year | 13 | 6
  Baseline: Missing | 0 | 0
  3 months: number analyzed (Participants) | 67 | 40
  3 months: Declined | 1 | 0
  3 months: Every month or so | 2 | 4
  3 months: Every week or more often | 16 | 9
  3 months: More than once a week | 8 | 2
  3 months: Never | 11 | 9
  3 months: Once or twice a month | 16 | 11
  3 months: Once or twice a year | 11 | 3
  3 months: Missing | 2 | 2
  6 months: number analyzed (Participants) | 67 | 41
  6 months: Declined | 0 | 1
  6 months: Every month or so | 5 | 6
  6 months: Every week or more often | 19 | 8
  6 months: More than once a week | 6 | 4
  6 months: Never | 12 | 6
  6 months: Once or twice a month | 13 | 8
  6 months: Once or twice a year | 10 | 8
  6 months: Missing | 2 | 0
  12 months: number analyzed (Participants) | 66 | 38
  12 months: Declined | 0 | 0
  12 months: Every month or so | 8 | 4
  12 months: Every week or more often | 18 | 8
  12 months: More than once a week | 5 | 5
  12 months: Never | 7 | 6
  12 months: Once or twice a month | 9 | 5
  12 months: Once or twice a year | 13 | 8
  12 months: Missing | 6 | 2

8. Other Pre Specified Outcome: Brief Multidimensional Measurement of Religiousness/Spirituality (BMMRS-adapted)
Description: Responses to "To what extent do you consider yourself a religious person? Responses ranged from "not religious at all" to "very religious." Higher scores indicated greater religiousness.
  Responses were used as a covariate in the initial Generalized linear mixed effect models.
  Prior research indicated that this item was associated with quality of life outcomes.
Time Frame: Change from baseline in religiousness/spirituality at 3, 6, and 12 months post baseline compared to controls
Population: Adolescents with cancer responses at baseline, 3, 6 and 12 months post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 83 | 43
Participants
  Baseline: Moderately religious | 34 | 22
  Baseline: Not religious at all | 16 | 6
  Baseline: Slightly religious | 23 | 9
  Baseline: Very religious | 10 | 6
  Baseline: Declined | 0 | 0
  Baseline: missing | 0 | 0
  3 months: number analyzed (Participants) | 67 | 40
  3 months: Moderately religious | 30 | 17
  3 months: Not religious at all | 15 | 7
  3 months: Slightly religious | 14 | 10
  3 months: Very religious | 6 | 4
  3 months: Declined | 0 | 0
  3 months: missing | 2 | 2
  6 months: number analyzed (Participants) | 67 | 41
  6 months: Moderately religious | 31 | 15
  6 months: Not religious at all | 18 | 6
  6 months: Slightly religious | 10 | 15
  6 months: Very religious | 5 | 4
  6 months: Declined | 1 | 1
  6 months: missing | 2 | 0
  12 months: number analyzed (Participants) | 66 | 38
  12 months: Moderately religious | 26 | 14
  12 months: Not religious at all | 15 | 8
  12 months: Slightly religious | 13 | 12
  12 months: Very religious | 6 | 2
  12 months: Declined | 1 | 0
  12 months: missing | 5 | 2

9. Other Pre Specified Outcome: Brief Multidimensional Measurement of Religiousness/Spirituality (BMMRS-adapted)
Description: Responses to "To What Extent do You Consider Yourself a spiritual person?" Responses ranged from "not spiritual at all" to "very spiritual." Higher score meant more spiritual. Reported are frequency distributions and percentages.
Time Frame: Baseline in religiousness/spirituality at 3, 6, and 12 months post-intervention. Used as a covariate in generalized linear mixed effect models.
Population: Adolescents with cancer responses at baseline, 3, 6 and 12 months post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 83 | 43
Participants
  Baseline: Moderately spiritual | 27 | 17
  Baseline: Not spiritual at all | 6 | 8
  Baseline: Slightly spiritual | 32 | 12
  Baseline: Very spiritual | 18 | 6
  Baseline: Declined | 0 | 0
  Baseline: Missing | 0 | 0
  3 months: number analyzed (Participants) | 67 | 40
  3 months: Moderately spiritual | 29 | 10
  3 months: Not spiritual at all | 8 | 5
  3 months: Slightly spiritual | 14 | 16
  3 months: Very spiritual | 14 | 7
  3 months: Declined | 0 | 0
  3 months: Missing | 2 | 2
  6 months: number analyzed (Participants) | 67 | 41
  6 months: Moderately spiritual | 23 | 11
  6 months: Not spiritual at all | 8 | 6
  6 months: Slightly spiritual | 24 | 19
  6 months: Very spiritual | 9 | 4
  6 months: Declined | 1 | 1
  6 months: Missing | 2 | 0
  12 months: number analyzed (Participants) | 66 | 38
  12 months: Moderately spiritual | 27 | 10
  12 months: Not spiritual at all | 8 | 7
  12 months: Slightly spiritual | 16 | 16
  12 months: Very spiritual | 8 | 3
  12 months: Declined | 2 | 0
  12 months: Missing | 5 | 2

10. Other Pre Specified Outcome: Brief Multidimensional Measurement of Religiousness/Spirituality (BMMRS-adapted)
Description: Responses to "How often do you pray privately?" Frequency of behavior was surveyed. Responses ranged from never to a few times a week. Higher scores indicated more praying privately.
  5 items were used in this study based on previous research with adolescent populations, which showed that these 5 items moderated study outcomes.
  Responses were used as covariates in the initial modeling.
Time Frame: Baseline in religiousness/spirituality at 3, 6, and 12 months post baseline compared to controls for adolescents only.
Population: Adolescents living with cancer Higher scores indicate increased frequency of experience or behavior. There are no missing data. The numbers analyzed in some rows differ from the Overall Number of Participants Analyzed for this Outcome Measure due either to missed study visits, attrition, or deaths at 3-months, 6-months, and 12-months.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 83 | 43
Participants
  How often do you pray privately?. Baseline.: A few times a month | 6 | 7
  How often do you pray privately?. Baseline.: A few times a week | 25 | 9
  How often do you pray privately?. Baseline.: Declined | 1 | 1
  How often do you pray privately?. Baseline.: Less than once a month | 6 | 3
  How often do you pray privately?. Baseline.: More than once a day | 9 | 7
  How often do you pray privately?. Baseline.: Never | 17 | 4
  How often do you pray privately?. Baseline.: Once a day | 11 | 10
  How often do you pray privately?. Baseline.: Once a month | 4 | 1
  How often do you pray privately?. Baseline.: Once a week | 4 | 1
  How often do you pray privately?. Baseline.: Missing | 0 | 0
  3 months.: number analyzed (Participants) | 67 | 40
  3 months.: A few times a month | 7 | 1
  3 months.: A few times a week | 15 | 5
  3 months.: Declined | 1 | 0
  3 months.: Less than once a month | 8 | 5
  3 months.: More than once a day | 8 | 6
  3 months.: Never | 10 | 6
  3 months.: Once a day | 10 | 11
  3 months.: Once a month | 1 | 2
  3 months.: Once a week | 5 | 2
  3 months.: Missing | 2 | 2
  How often do you pray privately. 6 months.: number analyzed (Participants) | 67 | 41
  How often do you pray privately. 6 months.: A few times a month | 5 | 3
  How often do you pray privately. 6 months.: A few times a week | 10 | 7
  How often do you pray privately. 6 months.: Declined | 1 | 1
  How often do you pray privately. 6 months.: Less than once a month | 6 | 3
  How often do you pray privately. 6 months.: More than once a day | 9 | 6
  How often do you pray privately. 6 months.: Never | 14 | 7
  How often do you pray privately. 6 months.: Once a day | 14 | 10
  How often do you pray privately. 6 months.: Once a month | 2 | 2
  How often do you pray privately. 6 months.: Once a week | 4 | 2
  How often do you pray privately. 6 months.: Missing | 2 | 0
  How often do you pray privately. 12 months.: number analyzed (Participants) | 66 | 38
  How often do you pray privately. 12 months.: A few times a month | 6 | 2
  How often do you pray privately. 12 months.: A few times a week | 10 | 7
  How often do you pray privately. 12 months.: Declined | 1 | 0
  How often do you pray privately. 12 months.: Less than once a month | 5 | 2
  How often do you pray privately. 12 months.: More than once a day | 11 | 6
  How often do you pray privately. 12 months.: Never | 11 | 8
  How often do you pray privately. 12 months.: Once a day | 11 | 5
  How often do you pray privately. 12 months.: Once a month | 3 | 2
  How often do you pray privately. 12 months.: Once a week | 3 | 4
  How often do you pray privately. 12 months.: Missing | 5 | 2

11. Other Pre Specified Outcome: Brief Multidimensional Measurement of Religiousness/Spirituality (BMMRS-adapted)
Description: Responses to item "I feel God's presence". Responses range from never to many times a day. Higher scores indicated greater experience of feeling God's presence.
  Prior research had demonstrated this item moderated study outcomes with respect to quality of life outcomes.
Time Frame: Baseline in religiousness/spirituality and at 3, 6, and 12 months post baseline compared to controls. Responses were used as a covariate in the initial generalized linear mixed effect models.
Population: Adolescents living with cancer.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 83 | 43
Participants
  Baseline: Declined | 2 | 2
  Baseline: Every day | 13 | 10
  Baseline: Many times a day | 10 | 6
  Baseline: Most days | 20 | 10
  Baseline: Never or almost never | 18 | 6
  Baseline: Once in a while | 11 | 7
  Baseline: Some days | 9 | 2
  Baseline: Missing | 0 | 0
  3 months: number analyzed (Participants) | 67 | 40
  3 months: Declined | 3 | 1
  3 months: Every day | 15 | 6
  3 months: Many times a day | 8 | 7
  3 months: Most days | 11 | 10
  3 months: Never or almost never | 9 | 4
  3 months: Once in a while | 9 | 5
  3 months: Some days | 10 | 5
  3 months: Missing | 2 | 2
  6 months: number analyzed (Participants) | 67 | 41
  6 months: Declined | 1 | 2
  6 months: Every day | 15 | 6
  6 months: Many times a day | 9 | 6
  6 months: Most days | 10 | 13
  6 months: Never or almost never | 10 | 5
  6 months: Once in a while | 11 | 5
  6 months: Some days | 9 | 4
  6 months: Missing | 2 | 0
  12 months: number analyzed (Participants) | 66 | 38
  12 months: Declined | 1 | 0
  12 months: Every day | 11 | 7
  12 months: Many times a day | 9 | 7
  12 months: Most days | 15 | 7
  12 months: Never or almost never | 12 | 6
  12 months: Once in a while | 4 | 6
  12 months: Some days | 9 | 3
  12 months: Missing | 5 | 2

12. Other Pre Specified Outcome: Satisfaction Questionnaire
Description: Items for this 13-item assessment of adolescent and family satisfaction with the FACE-TC intervention were developed using input from the community about the emotional of participation. Items are on a 5-point Likert scale from strongly disagree to strongly agree. 6 items were negative (felt afraid, too much to handle, harmful, angry, sad hurtful) and 7 items were positive (useful, helpful, load off my mind, satisfied, something I needed to do, courageous, worthwhile). Each subscale was scored separately. The minimum positive score was 17 and the maximum positive score was 35 for adolescents. The minimum negative score was 6 and the maximum negative score was 22 for adolescents. The minimum positive score was 11 and maximum score was 35 for family surrogate. The minimum negative score was 6 and the maximum negative score was 23 for surrogates. Higher score for positive scale was better outcome. Higher score for negative scale was worse outcome.
Time Frame: Two weeks post-baseline for control; two weeks post-baseline for intervention--immediately following Session 2. This was a process measure and as such is not reflected in the flow diagram, as it was not a primary or secondary outcome.
Population: Adolescents with cancer and their family surrogate decision makers responding agree or strongly agree to each item.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- FACE-TC Intervention: Participants (adolescents and family surrogate) randomized to the experimental condition receive Family Centered Advance Care Planning for Teens with Cancer (FACE-TC) intervention - 3 sessions scheduled one week apart of approximately 60 minutes duration each. Session 1 - Lyon Advance Care Planning Survey-Adolescent & Surrogate versions. Session 2 - Respecting Choices Interview facilitated by trained/certified facilitator with adolescent and family. Focuses on patient's understanding of their illness, possible complications, goals of care and treatment preferences in 3 bad outcome situations; and the Session 3 - Five Wishes an advance directive.
  FAmily CEntered Advance Care Planning for Teens with Cancer: 3 session weekly intervention: 1) survey completed by adolescent and family (surrogate decision maker) separately with facilitator; 2) Respecting Choices structured interview about patient's representation of illness, goals of care, hopes, treatment preferences; 3) completion of an advance directive.
- Treatment As Usual (TAU): Participants (adolescent/family dyads randomized to the treatment as usual (TAU) condition receive written information on advance care planning, but no active intervention.
Arm/Group | FACE-TC Intervention | Treatment As Usual (TAU)
Number analyzed (Participants) | 150 | 84
score on a scale
  Adolescents positive score: number analyzed (Participants) | 75 | 42
  Adolescents positive score | 26.8 (3.6) | 26.4 (3.8)
  Adolescent negative score: number analyzed (Participants) | 75 | 42
  Adolescent negative score | 11.2 (3.8) | 10.1 (3.2)
  Family surrogate positive score: number analyzed (Participants) | 75 | 42
  Family surrogate positive score | 28.1 (3.3) | 24.9 (4.4)
  Family surrogate negative score: number analyzed (Participants) | 75 | 42
  Family surrogate negative score | 11.4 (4.0) | 12.4 (4.1)
Statistical Analysis 1: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Adolescent positive score comparing intervention with TAU; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 0.72, Standard Error of Mean 0.71
Statistical Analysis 2: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Adolescent negative worded score comparing intervention to TAU; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.93, Standard Error of Mean 0.73
Statistical Analysis 3: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Family member positively worded score comparing intervention with treatment as usual; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 2.98, Standard Error of Mean 0.74
Statistical Analysis 4: Comparison: FACE-TC Intervention vs Treatment As Usual (TAU); Family member negative worded score comparing intervention to TAU; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -1.15, Standard Error of Mean 0.81

ADVERSE EVENTS:
Time Frame: From enrollment through study completion up to 18 months post-intervention (+/- 1 month study window).
Description: Potential adverse event data were collected over the 6 year trial period and reported in bi- annual to annual meetings with the Safety Monitoring Committee. Monthly investigator meetings consistently reviewed adverse events during the prior month and potential adverse events. Site monitoring visits also monitored adverse events and their documentation. All patients died from their cancer related illness or side effect of treatment. One parent died from disease progression of chronic illness.
Groups:
- FACE-TC Intervention Adolescent: Adolescent randomized with family member as dyad to the experimental condition receive Family Centered Advance Care Planning for Teens with Cancer (FACE-TC) intervention - 3 sessions scheduled one week apart of approximately 60 minutes duration each. Session 1 - Lyon Advance Care Planning Survey-Adolescent & Surrogate versions. Session 2 - Respecting Choices Interview facilitated by trained/certified facilitator with adolescent and family. Focuses on patient's understanding of their illness, possible complications, goals of care and treatment preferences in 3 bad outcome situations; and the Session 3 - Five Wishes an advance directive.
  FAmily CEntered Advance Care Planning for Teens with Cancer: 3 session weekly intervention: 1) survey completed by adolescent and family (surrogate decision maker) separately with facilitator; 2) Respecting Choices structured interview about patient's representation of illness, goals of care, hopes, treatment preferences; 3) completion of an advance directive.
- Treatment As Usual (TAU) Adolescent: Adolescent randomized with family member as dyad to the treatment as usual (TAU) condition receive written information on advance care planning, but no active intervention.
- FACE-TC Intervention Family Member: Family member randomized with adolescent as dyad to the experimental condition receive Family Centered Advance Care Planning for Teens with Cancer (FACE-TC) intervention - 3 sessions scheduled one week apart of approximately 60 minutes duration each. Session 1 - Lyon Advance Care Planning Survey-Adolescent & Surrogate versions. Session 2 - Respecting Choices Interview facilitated by trained/certified facilitator with adolescent and family. Focuses on patient's understanding of their illness, possible complications, goals of care and treatment preferences in 3 bad outcome situations; and the Session 3 - Five Wishes an advance directive.
  FAmily CEntered Advance Care Planning for Teens with Cancer: 3 session weekly intervention: 1) survey completed by adolescent and family (surrogate decision maker) separately with facilitator; 2) Respecting Choices structured interview about patient's representation of illness, goals of care, hopes, treatment preferences; 3) completion of an advance directive.
- TAU Family Member: Family member randomized with adolescent as dyad to the treatment as usual (TAU) condition receive written information on advance care planning, but no active intervention.
Arm/Group | FACE-TC Intervention Adolescent | Treatment As Usual (TAU) Adolescent | FACE-TC Intervention Family Member | TAU Family Member
All-Cause Mortality (participants affected / at risk) | 3/83 | 4/43 | 1/83 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/43 | 0/83 | 0/43
Other Adverse Events (participants affected / at risk) | 0/83 | 0/43 | 0/83 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT02693665/Prot_SAP_000.pdf
  • Informed Consent Form (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT02693665/ICF_001.pdf